CLINICAL TRIAL: NCT06996600
Title: Longitudinal Measurements of Flow in Cerebrospinal Fluid Shunts With a Wireless Thermal Anisotropy Measurement Device in People With Chronic Headaches
Brief Title: Assessment of CSF Shunt Flow and Headaches With a Thermal Measurement Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-01
Record Dates: First submitted 2025-05-12; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CSF Shunted Patients with Chronic Headaches (Experimental): hydrocephalus patients with an existing ventriculoperitoneal (VP) shunt who experience chronic headaches, defined as ≥15 headache episodes/month for ≥3 months
  Interventions: Device: wireless thermal anisotropy measurement device

INTERVENTIONS:
Device: wireless thermal anisotropy measurement device — Wireless wearable thermal anisotropy measurement device designed for use at home

SUMMARY:
This study evaluates the performance of a device for non-invasively assessing cerebrospinal fluid (CSF) shunt flow over multiple measurements performed by a study subject during headache and non-headache periods.

ELIGIBILITY:
Inclusion Criteria:

1. Existing ventriculoperitoneal CSF shunt
2. Subject experiencing ongoing headaches including at least 15 headache days per month for the past 3 months
3. Region of intact skin overlying an unambiguously identifiable palpable chronically indwelling ventricular shunt which crosses the clavicle and is appropriate in size for application of the study device
4. Available for remote and in-person follow-up during the 30-day measurement period
5. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
6. Subject or caregiver is able to clearly communicate and document information and shunt symptoms in English
7. Subject is at least 6 years old but not more than 80 years old

Exclusion Criteria:

1. Presence of more than one distal shunt catheter in the study device measurement region
2. Shunt is not palpable due to depth or depth of shunt where the device will be placed is greater than 4 mm per ultrasound evaluation
3. Presence of an interfering open wound or edema in the study device measurement region
4. Subject-reported history of serious adverse skin reactions to silicone-based adhesives
5. Investigator judges that the subject is likely to be lost to follow-up due to unavailability or clinical outcome being unobtainable
6. Investigator judges that the subject is unlikely to successfully take reliable measurements at home
7. Investigator judges that the subject/subject's caretaker would not be able to successfully place the device without assistance
8. Use of the study device would interfere with standard patient care, or emergency surgery that cannot be delayed, or participation in the study will interfere with, or be detrimental to, administration of optimal healthcare to the subject
9. Prior enrollment in this study
10. Participation in any other investigational procedural, pharmaceutical, and/or device study that may influence the collection of valid data under this study

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Study Device Flow Measurement and Subject-reported Headaches | 30 days
  Exploratory analysis to determine the relationship between headaches (subject-reported headache and non-headache periods) and measured flow. Data will be analyzed using the Point-Biserial Correlation Coefficient between headaches periods (headache and non-headache periods) and thermal flow score (flow score derived from algorithm analysis of raw thermal data)

CONTACTS AND LOCATIONS:
Locations (1):
- Rhaeos, Inc, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No